CLINICAL TRIAL: NCT06233604
Title: Dexamethasone vs. Dexmedetomidine for ESPB in Pain Management After Hip Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2/2024
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hip Osteoarthritis; Hip Arthropathy; Hip Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Sodium Chloride; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 0.2% ropivacaine for erector spinae plane block
  Interventions: Drug: 0.9%sodium chloride
- Dexamethasone (Experimental): 0.2% ropivacaine + 4mg Dexamethasone for erector spinae plane block
  Interventions: Drug: Dexamethasone
- Dexmedetomidine (Experimental): 0.2% ropivacaine + 50ug Dexmedetomidine for erector spinae plane block
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: 0.9%sodium chloride — unilateral administration of 20ml of 0,2% ropivacaine + 2ml 0.9% sodium chloride for the erector spine plane block
  Other Names: placebo
  Arms: Placebo
Drug: Dexamethasone — unilateral administration of 20ml of 0,2% ropivacaine with 4mg Dexamethasone for the erector spine plane block
  Arms: Dexamethasone
Drug: Dexmedetomidine — unilateral administration of 20ml of 0,2% ropivacaine with 50ug Dexmedetomidine for the erector spine plane block
  Arms: Dexmedetomidine

SUMMARY:
Effect of perineurial dexamethasone and dexmedetomidine on erector spinal plane block duration for hip arthroplasty

DETAILED DESCRIPTION:
This study is proposed to explore the effect of perineurial Dexamethasone and Dexmedetomidine on erector spinal plane block duration for spine surgery.

After spine surgery, patients need good analgesia. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anaesthesia is essential due to the much lower toxicity threshold of local anaesthetics. An effective adjuvant, such as Dexamethasone or Dexmedetomidine, could allow for a higher dilution of local anaesthetics while maintaining and enhancing their analgesic effect.

There is considerable research where intravenous and perineural dexamethasone and Dexmedetomidine use have been compared in adults. However, there is a massive lack of research regarding spine surgery and the Erector Spinae Plane Block.

In this study, investigators compare perineural Dexamethasone and Dexmedetomidine.

The investigator aims to find a dexamethasone or dexmedetomidine that covers the need for good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary hip arthroplasty
* aged >18 years and <100 years
* ASA physical status 1, 2 or 3.

Exclusion Criteria:

* if they refused to participate,
* had a history of opioid abuse,
* had an infection of the site of needle puncture,
* were less than 18 years of age,
* were postponed as having ASA 4 or 5,
* had an allergy to any of the drugs used in the study,
* renal failure (estimated glomerular filtration rate <15ml/min/1.73m2),
* liver failure,
* known or suspected coagulopathy,
* pre-existing anatomical or neurological disorders in the lower extremities,
* intellectual disability with problems in pain evaluation,
* severe psychiatric illness.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
first need of opiate | 48 hours after surgery
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid consumption | 48 hours after surgery
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 16 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 20 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
NLR | 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 48 hours after surgery
  Platelet-to-lymphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Wieczorowska-Tobis, Prof.dr hab., Study Chair — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No